CLINICAL TRIAL: NCT01964079
Title: The COMPAriSon of Systolic Blood Pressure Variability and Central Blood Pressure of Calcium Channel Blocker (Amlodipine) in Comparison With Angiotensin Receptor Blocker (Losartan) in Patients With Essential Hypertension
Brief Title: Comparision of Blood Pressure Variability Between Amlodipine and Losartan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Byung-Su Yoo, Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COMPASS-BPV
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CCB (amlodipine) (Active Comparator): For patients who fail to respond to 5 mg oral amlodipine daily, the dose will be titrated up to 10 mg amlodipineh. At subsequent visits, additional antihypertensive therapy (hydrochlorothiazide) will be added if systolic (>140 mmHg) or diastolic (>90 mmHg) BP is inadequate. Study drugs are administered once a day for 24 weeks. The dose will be titrated up if SBP is over 90 mmHg or there are no symptoms of hypotension (syncope, loss of consciousness, or orthostatic hypotension). If up-titration is not tolerable, because of side effects or hypotension, the previous dose will be administered as the final tolerable dose.
  Interventions: Drug: Amlodipine
- ARB (losartan) (Active Comparator): For patients who fail to respond to 50 mg oral losartan daily, the dose will be titrated up to 100 mg losartan. At subsequent visits, additional antihypertensive therapy (hydrochlorothiazide) will be added if systolic (>140 mmHg) or diastolic (>90 mmHg) BP is inadequate. Study drugs are administered once a day for 24 weeks. The dose will be titrated up if SBP is over 90 mmHg or there are no symptoms of hypotension (syncope, loss of consciousness, or orthostatic hypotension). If up-titration is not tolerable, because of side effects or hypotension, the previous dose will be administered as the final tolerable dose.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Amlodipine — Eligible subjects will be randomized 1:1 to either an amlodipine or a losartan group by a computer-generated random number table. For patients who fail to respond to 5 mg amlodipine, the dose will be titrated up to 10 mg amlodipine. At subsequent visits, additional antihypertensive therapy (hydrochlorothiazide) will be added if systolic (>140 mmHg) or diastolic (>90 mmHg) BP is inadequate. Study drugs are administered once a day for 24 weeks. The dose will be titrated up if SBP is over 90 mmHg or there are no symptoms of hypotension (syncope, loss of consciousness, or orthostatic hypotension). If up-titration is not tolerable, because of side effects or hypotension, the previous dose will be administered as the final tolerable dose.
  Other Names: Norvasc
  Arms: CCB (amlodipine)
Drug: Losartan — Eligible subjects will be randomized 1:1 to either an amlodipine or a losartan group by a computer-generated random number table. For patients who fail to respond to 50 mg losartan, the dose will be titrated up to 100 mg losartan. At subsequent visits, additional antihypertensive therapy (hydrochlorothiazide) will be added if systolic (>140 mmHg) or diastolic (>90 mmHg) BP is inadequate. Study drugs are administered once a day for 24 weeks. The dose will be titrated up if SBP is over 90 mmHg or there are no symptoms of hypotension (syncope, loss of consciousness, or orthostatic hypotension). If up-titration is not tolerable, because of side effects or hypotension, the previous dose will be administered as the final tolerable dose.
  Other Names: Cozaar
  Arms: ARB (losartan)

SUMMARY:
Blood pressure (BP) is believed to be a major determinant of vascular disease, and BP lowering is the most important goal in hypertension treatment. Thus, clinical guidelines for hypertension are mainly focused on lowering mean BP. However, despite an increasing incidence of stroke with age, the association between systolic BP (SBP) and the risk of stroke decreases with age. This disparity highlights a gap in the link between BP and vascular-related diseases (i.e., stroke). In clinical practice, visit-to-visit fluctuations in BP have been largely ignored and are thought to be an unreliable finding, even though this phenomenon is frequently observed. Rothwell et al. demonstrated that the visit-to-visit variability in SBP was a more powerful independent predictor of stroke than mean SBP, and that an increased residual variability in SBP in treated hypertensive patients was also a strong predictor of stroke and coronary events.

Recently updated (2011) hypertension guidelines from the National Institute for Health and Clinical Excellence (NICE) recommend an angiotensin converting enzyme inhibitor (ACEi) [or angiotensin II receptor blocker (ARB)] and calcium-channel blocker (CCB) as a first line drug. Although the significance of BP variability (BPV) has been illustrated, the main focus of the current guidelines is to reduce systolic and diastolic BP, not BPV.

In the X-CELLENT study, a CCB (amlodipine) and thiazide-like diuretic drug (indapamide sustained-release) led to a significant reduction in BPV, compared to an ARB (candesartan). In addition, the CCB showed the most effective reduction in systolic BPV among the antihypertensive drug class in a meta-analysis. However, there are no direct comparison studies of a CCB and ARB on BPV. Thus, we aim to compare the systolic BPV effects of a CCB versus an ARB in essential hypertensive patients. The primary hypothesis is that an ARB is not inferior to a CCB in the reduction of the systolic BPV standard deviation (SD) in essential hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older and below 80 years.
* Patients who have not previously taken any antihypertensive drugs or have discontinued previous antihypertensive drugs for 2 weeks.
* Mean SBP ≥140 mmHg or mean diastolic BP ≥ 90 mmHg (blood pressure will be checked at least 2 times in a seated position during the screening period).

Exclusion Criteria:

* Pregnant women, possible candidate for pregnancy, or breastfeeding women.
* Known or suspected secondary hypertension.
* Mean seated SBP ≥ 180 mmHg and/or mean seated diastolic BP ≥ 120 mmHg at any visit.
* Any clinically significant hepatic impairments.
* Severe renal impairment (serum creatinine level > 3.0 mg/dL or creatinine clearance < 30 mL/min).
* Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, or post-renal transplant.
* Clinically relevant hyperkalemia.
* Uncorrected volume or sodium depletion.
* Suspected primary aldosteronism.

  1. Hypertension and spontaneous or low-dose diuretic-induced hypokalemia.
  2. Drug-resistant hypertension, defined as sub-optimally controlled hypertension on a 3-drug program that includes an adrenergic inhibitor, vasodilator, and diuretic.
  3. Hypertension with adrenal incidentaloma.
  4. Hypertension and a family history of early-onset hypertension or cerebrovascular accident at a young age (<40 years).
  5. Hypertensive first-degree relatives of patients with primary aldosteronism.
* Symptomatic congestive heart failure.
* Angina pectoris requiring treatment.
* History of myocardial infarction or cerebrovascular accident (ischemic stroke or hemorrhage).
* History of refractory or potentially lethal arrhythmias.
* Concurrent participation in another clinical trial.
* Patients with known intolerance, contraindication, or hypersensitivity to any component of dihydropyridines or angiotensin II receptor blockers.
* Patients who are deemed unsuitable by the investigator.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
SD of visit-to-visit systolic blood pressure variability | 6 months
  Consecutive measured blood pressure values from each visit will be averaged, and the standard deviation (SD) is calculated using the mean systolic blood pressure of each visit.

SECONDARY OUTCOMES:
Central systolic blood pressure | 6 months
  Measurement of central blood pressure will be performed at randomization and 6 months.
Augmentation index of central blood pressure | 6 months
  Augmentation index of central blood pressure will be measured at randomization and 6 months.
Standard deviation of within-visit systolic blood pressure variability | 6 months
Coefficient of variation of visit-to-visit systolic blood pressure variability | 6 months
  The coefficient of variation (CV) is defined as the standard deviation/mean systolic blood pressure.
Variation independent of the mean of visit-to-visit systolic blood pressure variability | 6 months
  To eliminate the correlation of coefficient variation with mean SBP, we will calculate a further transformed variable, the variation independent of the mean (VIM). The VIM is defined as the standard deviation/mean^x, with x estimated from curve fitting of the data.
24-h ambulatory blood pressure monitoring | 6 months
Home systolic blood pressure | 6 months
  Home systolic blood pressure will be measured at each scheduled visit.

OTHER OUTCOMES:
Safety outcome | 6 months
  The number of all adverse events including laboratory tests, ECG changes, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Su Yoo, MD, PhD, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea